CLINICAL TRIAL: NCT02046122
Title: Safety and Efficacy of Chemotherapy Combined With Adoptive Transfer of Human Leukocyte Antigen (HLA)-Haploidentical Donor Lymphocyte Infusion (DLI) in Older Patients With Righ-Risk Acute Myeloid Leukemia (AML) and Myelodysplastic Syndrome (MDS)
Brief Title: Adoptive Transfer of Haplo-identical DLI for AML and MDS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00043247
Record Dates: First submitted 2014-01-23; First posted 2014-01-27 (Estimated); Results first posted 2018-07-18 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-12

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Idarubicin; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Idarubicin + Cytarabine + DLI (Experimental): Chemotherapy combined with adoptive transfer of HLA-haploidentical donor lymphocyte infusion (DLI)
  Interventions: Drug: Idarubicin; Drug: Cytarabine; Biological: DLI

INTERVENTIONS:
Drug: Idarubicin — Eligible subjects will receive induction chemotherapy with idarubicin (12 mg/m2 intravenously for 3 days) and cytarabine (100 mg/m2 intravenously for 7 days) starting Day 1 and ending Day 7. Patients 80 years or older will only receive 2 and 5 days of idarubicin and cytarabine respectively starting Day 1 and ending Day 5.
  Subjects who experience no remission or partial remission will receive a second course of the identical induction chemotherapy.
Drug: Cytarabine — Cytarabine (100 mg/m2 intravenously for 7 days) starting Day 1 and ending Day 7. Patients 80 years or older will only receive 2 and 5 days of idarubicin and cytarabine respectively starting Day 1 and ending Day 5.
  Subjects who achieve a complete remission (CR) will receive 2 further courses of cytarabine postremission chemotherapy (consolidation) at 1.0 g/m2 for 6 dosages followed by HLA-mismatched DLI after the second consolidation.
Biological: DLI — HLA-mismatched DLI will be administered Day 9, approximately 24-48 hours following completion of chemotherapy at a dose of 1x10^8 cluster of differentiation 3 (CD3+) cells; however, due to logistics of planning infusions with staffing, donor availability, weekends/holidays, etc., it may be necessary to postpone cell infusion up to 96 hours.
  Given the time constraints presented by the need to start induction chemotherapy as soon as possible, in some cases, it may not be logistically possible to administer cells with induction. In these cases, patients would just receive standard induction chemotherapy and cells would be administered after consolidation 1 in addition to consolidation 2
  Subjects who achieve a CR will receive 2 further courses of cytarabine postremission chemotherapy (consolidation) at 1.0 g/m2 for 6 dosages followed by HLA-mismatched DLI after the second consolidation.

SUMMARY:
The primary hypothesis is that chemotherapy followed by donor lymphocyte infusion (DLI) from HLA-haploidentical donors is a safe procedure that will not cause Graft versus Host Disease (GVHD) or increased treatment-related mortality. The Investigator further believes that this will improve outcomes of elderly patients with high-risk AML or MDS compared to chemotherapy alone, and that that this benefit will be even greater in donor-recipient pairs that share maternal-fetal microchimerism or non-inherited maternal antigen (NIMA) mismatch. A large part of this trial will include immune function assays as well as assessments of efficacy, toxicity, and GVHD. Because this therapy may be a tolerable alternative to allogeneic hematopoietic stem cell transplantation (alloHSCT) for elderly patients, the Investigator will validate functional measurements (e.g. Comprehensive Geriatric Assessment (CGA)) with biologic correlates (cytokine and genomic profiles) and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have their diagnosis of high-risk AML or high-risk MDS confirmed by pathologic review of bone marrow biopsy according to WHO guidelines
2. Patients will be defined as high risk AML and thus eligible if they meet one or more of the following criteria:

   1. Secondary AML (from underlying MDS or therapy related)
   2. Presence of complex cytogenetic abnormalities (3 or more cytogenetic abnormalities), all monosomies, del 5q, del 7q, inv3, t(3;3), t(6;9), t(9;22), abn 11q23 (excluding t(9;11))
   3. Fms-like tyrosine kinase 3 (FLT3)-internal tandem duplication (ITD) mutation positive
   4. Age ≥ 65 years given poor outcomes even with favorable cytogenetics
3. Patients will be defined as high risk MDS and thus eligible if they have a MD Anderson Comprehensive Cancer MDS Risk Score ≥9
4. Subjects must have Eastern Cooperative Oncology Group (ECOG) Performance status of 0,1,or 2; if ECOG 2, they must also have a Charlson comorbidity index of ≤5.
5. Subjects must be 55 years of age or older
6. Subjects should have a 3-5/6 HLA-matched related haploidentical donor who is evaluated and deemed able to provide DLI.
7. Patient should be able to provide informed consent
8. Subjects must have a multigated acquisition (MUGA) and /or ECHO or cardiac magnetic resonance imaging (MRI). The required minimum standards include MUGA or ECHO or cardiac MR showing an ejection fraction( EF) of 40%. Those with an EF 40-49% must also have a cardiologist consult and assist with management.
9. Pulmonary function tests (PFTs) with diffusing capacity of lung for carbon monoxide (DLCO) are conditional for subjects at the discretion of the physician. The required minimum standards for those who have PFTs include DLCO of 40%. Those with DLCO of 40-49% must have a pulmonologist consult and assist with management.
10. Subjects of all genders and races are eligible

Exclusion Criteria:

1. Pregnant or lactating women.
2. Patients with other major medical or psychiatric illnesses which the treating physician feels could seriously compromise tolerance to this protocol
3. Patients with known active central nervous system (CNS) disease
4. Patients with acute promyelocytic leukemia (FAB M3)

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-07; Primary Completion 2017-06-15 (Actual); Study Completion 2019-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Sung, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 subject was a screen failure and 1 subject withdrew prior to starting study.
Groups:
- Idarubicin + Cytarabine + DLI: Chemotherapy combined with adoptive transfer of HLA-haploidentical donor lymphocyte infusion (DLI)
  Idarubicin: Eligible subjects will receive induction chemotherapy with idarubicin (12 mg/m2 intravenously for 3 days) and cytarabine (100 mg/m2 intravenously for 7 days) starting Day 1 and ending Day 7. Patients 80 years or older will only receive 2 and 5 days of idarubicin and cytarabine respectively starting Day 1 and ending Day 5.
  Subjects who experience no remission or partial remission will receive a second course of the identical induction chemotherapy.
  Cytarabine: Cytarabine (100 mg/m2 intravenously for 7 days) starting Day 1 and ending Day 7. Patients 80 years or older will only receive 2 and 5 days of idarubicin and cytarabine respectively starting Day 1 and ending Day 5.
  Subjects who achieve a complete remission (CR) will receive 2 further courses of cytarabine postremission chemotherapy (consolidation) at 1.0 g/m2 for 6 dosages followed by HLA-mismatched DLI after
Period: Overall Study
Arm/Group | Idarubicin + Cytarabine + DLI
Started | 17
Completed | 8
Not Completed | 9
Not completed — Physician Decision | 8
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Overall Number of Baseline Participants represents the number of participants who were Enrolled.
Arm/Group | Idarubicin + Cytarabine + DLI
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 71 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 15
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Unacceptable Toxicity
Description: Unacceptable toxicity is defined as:
  i. Grade III or IV acute GVHD (aGVHD) of the gut or liver or Grade IV aGVHD of the skin lasting > 7 days;
  ii. Grade IV Common Terminology Criteria for Adverse Events (CTCAE) toxicity attributable to DLI (e.g. infusion reaction, as opposed to Grade IV CTCAE toxicity from chemotherapy) and lasting >7 days
  iii. Treatment-related mortality (TRM)
Time Frame: up to 8 weeks after last cell infusion
Measure: Count of Participants; unit: Participants
Arm/Group | Idarubicin + Cytarabine + DLI
Number analyzed (Participants) | 17
Participants | 1

2. Secondary Outcome: Disease Free Survival
Description: 1 year disease free survival rate following adoptive transfer
Time Frame: one year following adoptive transfer
Population: Data not collected on one subject.
Measure: Count of Participants; unit: Participants
Arm/Group | Idarubicin + Cytarabine + DLI
Number analyzed (Participants) | 16
Participants | 3

3. Secondary Outcome: Overall Survival
Description: Number of participants alive 2 years after completing adoptive transfer therapy.
Time Frame: 2 years after completing therapy
Population: Seventeen patients were enrolled between 2014 and 2017 with a median follow-up time of 299 days among all patients. One enrolled patient who developed sepsis during induction chemotherapy did not receive MST, and was excluded from final analysis of safety and efficacy.
Measure: Number; unit: participants
Arm/Group | Idarubicin + Cytarabine + DLI
Number analyzed (Participants) | 16
participants | 16

4. Secondary Outcome: Percentage of Subjects With Acute GVHD
Description: Grade III or IV aGVHD of the gut or liver or Grade IV aGVHD of the skin lasting > 7 days
Time Frame: 8 weeks after last cell infusion
Measure: Number; unit: percentage of participants
Arm/Group | Idarubicin + Cytarabine + DLI
Number analyzed (Participants) | 17
percentage of participants | 0

5. Secondary Outcome: Percentage of Subjects With Unacceptable Toxicity
Description: Grade IV CTCAE toxicity attributable to DLI (e.g. infusion reaction, as opposed to Grade IV CTCAE toxicity from chemotherapy) and lasting >7 days, Grade III or IV aGVHD of the gut or liver or Grade IV aGVHD of the skin lasting > 7 days, or death
Time Frame: 8 weeks after the last cell infusion
Measure: Number; unit: percentage of participants
Arm/Group | Idarubicin + Cytarabine + DLI
Number analyzed (Participants) | 17
percentage of participants | 5.88

6. Secondary Outcome: Rate of Efficacy
Description: Efficacy as measured by the number of subjects with a complete remission. Responses were evaluated according to standard criteria defined by the National Comprehensive Cancer Network Guidelines for AML (www.nccn.org).
Time Frame: 2 years after completing therapy
Population: Data not collected on one subject.
Measure: Count of Participants; unit: Participants
Arm/Group | Idarubicin + Cytarabine + DLI
Number analyzed (Participants) | 16
Participants | 10

7. Secondary Outcome: Number of Participants With Immune Recovery
Description: Immune recovery determined by measurements of cytokine profiles, lymphocyte and natural killer (NK) enumeration and flow-based assays, measured prior to induction, prior to each round of consolidation, 8 weeks after the last cycle of consolidation, and every 3 months after treatment for up to 2 years
Time Frame: up to 2 years after completing therapy
Population: Data not collected on one subject.
Measure: Count of Participants; unit: Participants
Arm/Group | Idarubicin + Cytarabine + DLI
Number analyzed (Participants) | 16
Participants | 3

8. Secondary Outcome: Number of Days to Hematopoietic Recovery
Description: Hematopoietic recovery as measured by the date of the first of three consecutive laboratory values where the absolute neutrophil count (ANC) ≥ 500/μl , the date of the first of three consecutive laboratory values obtained on different days where the platelet count was > 20,000/μl without transfusion.
Time Frame: 2 years after completion of therapy
Population: Data not collected on one subject.
Measure: Median (Full Range); unit: days
Arm/Group | Idarubicin + Cytarabine + DLI
Number analyzed (Participants) | 16
days
  Neutrophil recovery | 29 [16 to 31]
  Platelet recovery | 32 [23 to 37]

ADVERSE EVENTS:
Time Frame: All serious adverse events (SAEs) that occur up to 30 days after the last Donor Lymphocyte Infusion (DLI) will be reported.
Description: After 30 days, SAEs will be reported if thought related to treatment for the duration of the study. Non-treatment related SAEs were not collected past 30 days after the last DLI.
Arm/Group | Idarubicin + Cytarabine + DLI
All-Cause Mortality (participants affected / at risk) | 12/17
Serious Adverse Events (participants affected / at risk) | 8/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Idarubicin + Cytarabine + DLI (N=17)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Multi-organ failure (General disorders) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Idarubicin + Cytarabine + DLI (N=17)
Anemia (Blood and lymphatic system disorders) | 13 (65)
Blood and lymphatic system disorders other (Blood and lymphatic system disorders) | 4 (7)
Febrile neutropenia (Blood and lymphatic system disorders) | 13 (21)
Atrial fibrillation (Cardiac disorders) | 1 (1)
cardiac disorders other (Cardiac disorders) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 1 (1)
eye disorders other (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 3 (3)
Fever (Infections and infestations) | 1 (1)
general disorders and administration site conditions (Infections and infestations) | 1 (1)
Infections and infestations other (Infections and infestations) | 2 (2)
Lung infection (Infections and infestations) | 1 (1)
Penile infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 6 (6)
Splenic infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3)
Blood bilirubin increased (Investigations) | 2 (2)
Creatinine increased (Investigations) | 1 (1)
ECG QT corrected interval prolonged (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (2)
Neutrophil count decreased (Investigations) | 11 (16)
Platelet count decreased (Investigations) | 17 (34)
White blood cell decreased (Investigations) | 16 (28)
Acidosis (Metabolism and nutrition disorders) | 1 (2)
Alkalosis (Metabolism and nutrition disorders) | 1 (3)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 7 (18)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 7 (8)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 11 (26)
Hyponatremia (Metabolism and nutrition disorders) | 2 (4)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders other (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 3 (4)
Hypotension (Vascular disorders) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-07-10): https://cdn.clinicaltrials.gov/large-docs/22/NCT02046122/Prot_SAP_000.pdf
  • Informed Consent Form (2018-01-04): https://cdn.clinicaltrials.gov/large-docs/22/NCT02046122/ICF_001.pdf